CLINICAL TRIAL: NCT07122375
Title: Reliability and Normative Results of Angle-Specific Torque Profile Analysis in the Wrist Joint
Brief Title: Angle-Specific Torque Profile Analysis in the Wrist Joint
Status: Not yet recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Barış SEVEN, Principal Investigator, Assistant Professor, Gazi University
Other Study IDs: 9
Record Dates: First submitted 2025-07-30; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Wrist; Reliability; Torque; Isokinetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Angle Specific Torque Profile Analysis — All assessment data will be obtained from the archival records of young healthy adults, and no new assessments will be conducted. Raw data from wrist flexion and extension evaluations performed using an isokinetic dynamometer will be utilized.

SUMMARY:
The wrist joint performs various tasks at multiple angles during daily activities, both in flexion and extension positions. Among the parameters that facilitate these tasks, strength-particularly in relation to coordination and motor control-plays a key role. Therefore, identifying potential strength deficits is important for maintaining the continuity of daily functional tasks. In the literature, a wide range of methods exist for evaluating strength, from manual tests to advanced technological devices (references). One such method, isokinetic dynamometry, is considered among the most reliable due to its ability to provide objective and standardized measurements across different types of muscle contractions (isometric, isotonic, and isokinetic). Isokinetic dynamometers yield various data including peak torque, average torque, total work, fatigue index, and torque slope. Researchers frequently interpret findings based on peak or average torque values generated during isokinetic contractions. These torque measures provide an overall representation of strength during a given movement.

In wrist movements, rather than a single muscle, muscle groups are responsible for executing motion. However, when only peak or average torque at a single joint angle is assessed, the presence or absence of weakness in the movement can be detected, but it offers limited information. If weakness exists, identifying the specific joint angle at which it occurs can provide more direct insights into which muscles may be impaired. Furthermore, angle-specific profiling allows for characterization of muscle behavior throughout the movement, offering valuable information about potential kinematic disruptions. Having normative data on these profiles enables the detection of deviations from typical patterns across the full range of motion, which can be beneficial for both diagnosis and treatment planning.

However, to derive such benefits, it is critical that the data be obtained using reliable methods. Reliability refers to the degree to which an instrument or technique yields consistent results across repeated measurements, and is a prerequisite for usability. Statistical Parametric Mapping (SPM) is an increasingly popular method that enables angle-specific torque analysis, providing clinically and scientifically meaningful information on muscle strength. Angle-specific mapping is considered the "gold standard" because it presents torque values across the entire joint range, eliminating the need for interpolation between angles. For example, during daily activities, the wrist joint commonly operates within a range from 40° extension to 38° flexion. Therefore, measuring strength at only one joint angle may not be sufficient to reflect the potential limitations experienced in everyday tasks.

Despite its advantages, no reliability study involving SPM analysis has been found for the wrist joint. Furthermore, there is currently no study providing normative data for SPM-based analysis in the wrist. The aim of this study is to examine the reliability of angle-specific torque profile analysis during wrist flexion and extension movements and to provide normative data for healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adult participants

Exclusion Criteria:

* Participants who were unable to complete the target range of motion
* Participants with missing data

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adult participants
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Angle Specific Torque Profile Analysis | 4 months
  Raw data from the system files of the isokinetic dynamometer of both extremities of the participants who meet the criteria will be collected. SPM analysis of these raw data will be performed using the open source spm1d package in Matlab (R2021b, The Mathworks Inc, Natick, MA) software. Thus, the torque/angle data generated by the movements of both extremities through the range of motion set in the isokinetic dynamometer will be divided into 101 slices and angle-dependent torque graphs will be generated (SPM analysis). SPM analysis will be performed for wrist flexors and extensors. As a result of this analysis, the angle-dependent torque characteristics of both wrists and unilateral angle-dependent agonist/antagonist torque characteristics will be examined.

IPD SHARING:
Plan to Share IPD: Undecided